CLINICAL TRIAL: NCT02152332
Title: A Randomized, Double-blind, Placebo- and Positive-controlled, Multiple-dose, Four-way, Cross-over Study to Evaluate the Effects of Repeated Oral Doses of JNJ-54861911 on Electrocardiogram Intervals in Healthy Subjects
Brief Title: A Study to Evaluate the Effects of JNJ-54861911 on Electrocardiogram Intervals in Healthy Particiants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR104508; 54861911ALZ1007 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: JNJ-54861912; RSC-385896; MTS-0385896A; Phase 1; Moxifloxacin; Placebo; Healthy
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment Sequence Group ADBC (Experimental): Participant will receive Treatment A (JNJ-54861911, 50 milligram (mg) once daily for 7 days plus moxifloxacin-matched placebo on Day 7) followed by Treatment D (JNJ-54861911-matched placebo once daily for next 7 days plus moxifloxacin 400 mg on Day 7 of second treatment regimen, then Treatment B (JNJ-54861911, 150 mg once daily for next 7 days plus moxifloxacin-matched placebo on Day 7 of third treatment regimen followed by Treatment C (JNJ-54861911-matched placebo once daily for next 7 days plus moxifloxacin-matched placebo on Day 7 of fourth treatment regimen).
  Interventions: Drug: JNJ-54861911-Therapeutic Dose; Drug: JNJ-54861911 - Supratherapeutic Dose; Drug: JNJ-54861911-Matched Placebo; Drug: Moxifloxacin; Drug: Moxifloxacin Matched Placebo
- Treatment Sequence Group BACD (Experimental): Participant will receive Treatment B (JNJ-54861911, 150 mg once daily for 7 days plus moxifloxacin-matched placebo on Day 7) followed by Treatment A (JNJ-54861911, 50 mg once daily for next 7 days plus moxifloxacin-matched placebo on Day 7 of second treatment regimen), then Treatment C (JNJ-54861911-matched placebo once daily for next 7 days plus moxifloxacin-matched placebo on Day 7 of third treatment regimen) followed by followed by Treatment D (JNJ-54861911-matched placebo once daily for next 7 days plus moxifloxacin 400 mg on Day 7 of fourth treatment regimen).
  Interventions: Drug: JNJ-54861911-Therapeutic Dose; Drug: JNJ-54861911 - Supratherapeutic Dose; Drug: JNJ-54861911-Matched Placebo; Drug: Moxifloxacin; Drug: Moxifloxacin Matched Placebo
- Treatment Sequence Group CBDA (Experimental): Participant will receive Treatment C (JNJ-54861911-matched placebo once daily for next 7 days plus moxifloxacin-matched placebo on Day 7) followed by Treatment B (JNJ-54861911, 150 mg once daily for next 7 days plus moxifloxacin-matched placebo on Day 7 on second treatment regimen), then Treatment D (JNJ-54861911-matched placebo once daily for next 7 days plus moxifloxacin 400 mg on Day 7 of third treatment regimen) followed by Treatment A (JNJ-54861911, 50 mg once daily for next 7 days plus moxifloxacin-matched placebo on Day 7 of fourth treatment regimen).
  Interventions: Drug: JNJ-54861911-Therapeutic Dose; Drug: JNJ-54861911 - Supratherapeutic Dose; Drug: JNJ-54861911-Matched Placebo; Drug: Moxifloxacin; Drug: Moxifloxacin Matched Placebo
- Treatment Sequence Group DCAB (Experimental): Participant will receive Treatment D (JNJ-54861911-matched placebo once daily for 7 days plus moxifloxacin 400 mg on Day 7) followed by Treatment C (JNJ-54861911-matched placebo once daily for next 7 days plus moxifloxacin-matched placebo on Day 7 of second treatment regimen), then Treatment A (JNJ-54861911, 50 mg once daily for next 7 days plus moxifloxacin-matched placebo on Day 7 of third treatment regimen) followed by Treatment B (JNJ-54861911, 150 mg once daily for next 7 days plus moxifloxacin-matched placebo on Day 7 on fourth treatment regimen).
  Interventions: Drug: JNJ-54861911-Therapeutic Dose; Drug: JNJ-54861911 - Supratherapeutic Dose; Drug: JNJ-54861911-Matched Placebo; Drug: Moxifloxacin; Drug: Moxifloxacin Matched Placebo

INTERVENTIONS:
Drug: JNJ-54861911-Therapeutic Dose — JNJ-54861911 50 mg once daily for 7 days in all treatment sequence.
  Other Names: RSC-385896; MTS-0385896A
Drug: JNJ-54861911 - Supratherapeutic Dose — JNJ-54861911 150 mg once daily for 7 days in all treatment sequence.
  Other Names: RSC-385896; MTS-0385896A
Drug: JNJ-54861911-Matched Placebo — JNJ-54861911-matched placebo once daily for 7 days in all treatment sequence.
Drug: Moxifloxacin — Moxifloxacin 400 mg on Day 7 in all treatment sequence.
Drug: Moxifloxacin Matched Placebo — Moxifloxacin matched placebo, 400 mg on Day 7 in all treatment sequence.

SUMMARY:
The purpose of this study is to evaluate the effects of JNJ-54861911 on the QT/QTc intervals in healthy participants, when administered at therapeutic (50 milligram [mg] once-daily) and supratherapeutic (150 mg once-daily) doses for 7 days.

DETAILED DESCRIPTION:
This is a Phase 1, double blind (a medical research study in which neither the researchers nor the participants know what treatment the participants is receiving), randomized (study drug assigned by chance), placebo and positive-controlled, multiple-dose, 4-way crossover (method used to switch participants from one study group to another) study. The study consists of 3 parts: Screening period (Days -21 to -2), Double-blind treatment period and End-of-study/early withdrawal assessment period (9 to 13 days after last dose). Treatment period will comprise of 4 treatment regimens each consisting of a baseline assessment and a treatment regime (Days -1 to 9). The participants will be randomly assigned to 1 of 4 treatment sequence groups (ADBC, BACD, CBDA, and DCAB) based on a computer-generated randomization schedule and will receive the following 4 treatments in the order specified by the randomization: Treatment A (JNJ-54861911, 50 milligram (mg) once daily for 7 days plus moxifloxacin-matched placebo on Day 7); Treatment B (JNJ-54861911, 150 mg once daily for 7 days plus moxifloxacin-matched placebo on Day 7); Treatment C (JNJ-54861911-matched placebo once daily for 7 days plus moxifloxacin-matched placebo on Day 7); Treatment D (JNJ-54861911-matched placebo once daily for 7 days plus moxifloxacin 400 mg on Day 7). Each treatment period will be separated by a washout period of at least 6 - 10 days. Total duration of study for a participant will be 93 days. Change from Baseline in QT/QTc intervals at Day 7 will be evaluated as primary end point. Participant's safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent document indicating they understand the purpose of and procedures required for the study, including the required pharmacogenomics component (which specifies testing of genes predisposing to long or short QT and related cardiac syndromes), and are willing to participate in the study
* If a woman, must be either a) Not of childbearing potential: postmenopausal (greater than [>] 45 years of age with amenorrhea for at least 2 years, or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone [FSH] >40 international units per milliliter [IU/mL])or surgically sterile; b) Of child-bearing potential and be practicing an effective method of birth control
* If a man, who is sexually active with a woman of child-bearing potential and has not had a vasectomy, must agree to use an adequate contraception method as deemed appropriate by the investigator
* An average of triplicate 12-lead electrocardiogram (ECG) recordings, completed within 4 minutes total, consistent with normal cardiac conduction and function, including: a) normal sinus rhythm with heart rate between 45 and 100 beats per minutes (inclusive); b) QTcF interval between 350 to 450 milliseconds, inclusive; c) QRS interval of less than (<) 110 milliseconds; d) PR interval <200 milliseconds; e) PR interval <200 milliseconds; f) ECG morphology consistent with healthy cardiac conduction and function
* Blood pressure (after the participants remains supine for 5 minutes) between 90 and 140 milimeters of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, gastro-intestinal disease, or any other illness that the investigator considers should exclude the parrticipants or that could interfere with the interpretation of the study results
* History of additional risk factors for torsade de pointes or the presence of a family history of Short QT Syndrome, Long QT Syndrome, abnormal bleeding or blood clotting, sudden unexplained death at a young age (less than/equal to 40 years), drowning or sudden infant death syndrome in a first degree relative (that is, biological parent, sibling, or child)
* Use of any prescription medication (with the exception of hormonal contraceptives or hormonal replacement therapy) within 14 days before Day -1 of Period 1; use of nonprescription medication (including vitamins and herbal supplements such as St. John's Wort) except for acetaminophen, within 30 days before Day -1 of Period 1; acetaminophen within 3 days of study drug administration in each treatment period
* Clinically significant abnormal values for hematology, clinical chemistry (including hypo- or hyperkalemia, -magnesemia, or -calcemia) or urinalysis at Screening or at admission to the study center for Period 1 as deemed appropriate by the Investigator
* Clinically significant abnormal physical examination, vital signs or 12-lead ECG at Screening or at admission to the study center for Period 1 as deemed appropriate by the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in QT/QTc interval at Day 7 | Baseline and Day 7

SECONDARY OUTCOMES:
Change From Baseline in Other Electrocardiogram (ECG) Parameters at Day 7 | Baseline and Day 7
  Other ECG parameters included RR interval, PR interval and QRS interval.
Maximum Plasma Concentration (C[max]ss) at Steady State | Pre-dose and 3 hour (hr) post dose on Day 1, 3, 5, and 7; 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, 12, 16, 24 hrs post dose on Day 7
  The C(max)ss is the maximum plasma concentration at steady state which will be observed during dosing interval.
Minimum Plasma Concentration (C[min]ss) at Steady State | Pre-dose and 3 hour (hr) post dose on Day 1, 3, 5, and 7; 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, 12, 16, 24 hrs post dose on Day 7
  The C(min)ss is the minimum plasma concentration at steady state which will be observed during dosing interval.
Trough Plasma Concentration (C[trough]) | Pre-dose and 3 hour (hr) post dose on Day 1, 3, 5, and 7; 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, 12, 16, 24 hrs post dose on Day 7
  Trough plasma concentration is the plasma concentration before dosing or at the end of the dosing interval of any dose other than the first dose.
Time to Reach the Maximum Plasma Concentration (T[max]) | Pre-dose and 3 hour (hr) post dose on Day 1, 3, 5, and 7; 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, 12, 16, 24 hrs post dose on Day 7
  The T[max] is time to reach the observed maximum plasma concentration.
Average Plasma Concentration at Steady State (C[avg]ss) | Pre-dose and 3 hour (hr) post dose on Day 1, 3, 5, and 7; 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, 12, 16, 24 hrs post dose on Day 7
  Average Plasma Concentration at Steady State (C[avg]ss) will be calculated as Area under the plasma concentration-time curve (AUC[tau]) divided by the dosing interval (tau).
Area Under the Plasma Concentration-Time Curve During a Dosing Interval (AUC[tau]ss) | Pre-dose and 3 hour (hr) post dose on Day 1, 3, 5, and 7; 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, 12, 16, 24 hrs post dose on Day 7
  The AUC ([tau]ss) is the area under the plasma concentration time curve observed during a dosing interval.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trials, Study Director — Janssen Research & Development, LLC
Locations (1):
- Tempe, Arizona, United States